CLINICAL TRIAL: NCT01183793
Title: MR Enterography Assessment of Post Operative Small Bowel Length in Short Bowel Syndrome Patients
Brief Title: Magnetic Resonance (MR) Enterography Assessment of Post Operative Small Bowel Length in Short Bowel Syndrome Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Departement de la Recherche Clinique et de l'Innovation, CHU de NICE
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 09-CIR-02
Record Dates: First submitted 2010-08-02; First posted 2010-08-18 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2010-06

CONDITIONS: Short Bowel Syndrome
Keywords: Gastrointestinal Tract [A03.556]
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bras pair (Other): MR-enterography then barium follow through
  Interventions: Radiation: Barium follow-through and MR-enterography
- Bras impair (Other): Barium follow-through then MR-enterography
  Interventions: Radiation: Barium follow-through and MR-enterography

INTERVENTIONS:
Radiation: Barium follow-through and MR-enterography — Assessment of the lack of difference between surgical and MR enterography small bowel length measurement with a comparison sample test

SUMMARY:
It is essential to know intestinal length and anastomotic type in post-operative short bowel syndrome patients. These parameters can help predict long-term intestinal failure with long-term parenteral nutrition usually needed for smallest lengths. Sometimes these parameters are unfortunately missing for lack of intraoperative measurement. Thus, it is necessary to develop non-invasive and reproducible techniques to assess small bowel length. This is the reason why the investigators will evaluate magnetic resonance (MR)-enterography and barium follow-through in this indication. There are at this time only two small studies evaluating barium follow-through for intestinal length measurement, and none evaluating MR-enterography. However, a major advantage of the latter is the lack of radiation exposure and possibility to perform 3D.

This will be an open labelled single center crossover study. Short bowel syndrome patients of the investigators center will be included after consent. The sequence of exams (MR enterography followed by barium follow-through or vice-versa) will be randomly assigned. Peroperative short bowel length measurement will be available for all patients. There will be one month between the two exams.

The main objective of this study is to assess the performance of MR-enterography in short bowel measurement in short bowel syndrome patients, the gold standard being peroperative length. Secondary objectives are to assess the performance of barium follow-through in short bowel measurement in these patients, and to show that barium follow-through does not perform better than MR-enterography. For that purpose the investigators will include 50 patients over 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Intraoperative small bowel length < 200 cm
* Males and females between 18 and 85 years of age
* Patient with social insurance
* Signature of informed consent

Exclusion Criteria:

* Allergy to contrast product
* Enterostomy closure expected within 2 months after randomization
* Pregnancy or breast feeding woman
* Swallowing disorders
* Deprivation of liberty
* Contraindications to magnetic resonance imaging (pace-maker, metal implant, known allergy to gadolinium)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-10 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of the lack of difference between surgical and MR enterography small bowel length measurement with a comparison sample test | at 3 months

SECONDARY OUTCOMES:
Assessment of the lack of difference between surgical and barium follow through small bowel length measurement with a comparison sample test | at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: SCHNEIDER Stephane, PU-PH, Principal Investigator — Services d'Hépato-Gastroentérologie et Nutrition Clinique
Locations (1):
- Service d'Hépato-Gastroentérologie et Nutrition Clinique - CHU Nice - hôpital Archet 2, Nice, France